CLINICAL TRIAL: NCT01163513
Title: Cardiovascular Disease Research Using Linked Bespoke Studies and Electronic Records
Brief Title: Coronary Mortality in South Asians: Aetiologic and Prognostic Effects
Acronym: CALIBER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: DR M. JUSTIN ZAMAN, University College, London
Other Study IDs: CALIBER 09-01
Record Dates: First submitted 2010-04-16; First posted 2010-07-15 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2010-07

CONDITIONS: Acute Coronary Syndromes
Keywords: ethnicity; prognosis
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- White population
- Indian
- Pakistani
- Bangladeshi
- Other: other South Asian

SUMMARY:
The purpose of this study is to determine the extent to which South Asian ethnicity is both an etiologic and prognostic factor for coronary disease, and investigate factors influencing outcomes.

DETAILED DESCRIPTION:
Coronary death rates among first-generation migrants from South Asia are higher than those of the White majority population. Understanding the relative contribution of incidence and case fatality to overall coronary death rates allows preventive interventions to be targeted where they are likely to be more efficacious.

We seek to do this by meta-analysing new data with previously published work identified after systematic review of published literature. We will combine studies spanning different modes of presentation with coronary disease from 'normal' populations to suspected stable angina to higher-risk patients diagnosed with ACS within a national registry [MINAP].

Initially we will undertake retrospective cohort studies using four new databases (The aetiologic healthy population study, the Whitehall II Study; The chest pain clinic cohort with new-onset chest pain; the coronary angiography cohort (ACRE) and an acute coronary syndrome cohort, the Myocardial Infarction National Audit Project (MINAP).

We will define ethnicity according to the UK Office for National Statistics 1991 census categories. All four cohorts are flagged for mortality with the Office for National Statistics.

We will use a combined non-fatal outcome (non-fatal myocardial infarction and admission with angina) in the aetiologic cohort, as well as risk of coronary death. We will assess risk of coronary death in the chest pain clinic and coronary angiogram cohorts and all-cause death in the acute coronary syndrome cohort as cause-specific death is unavailable. We will assess prognosis for coronary death in Whitehall-II among those who had had typical angina at baseline. We will perform Cox proportional hazards regression adjusted for age (as a continuous variable), sex, hypertension, blood cholesterol, smoking and diabetes in all cohorts. We will then stratify these analyses in our prognostic studies by age, diabetes, ACS type, deprivation, smoking and secondary prevention management and formally examine whether a statistical difference exists between the hazard ratio of strata with the Bland-Altman two-tailed test of interaction.

We will combine results of new and older studies and calculate pooled odds ratios, weights, and 95% confidence intervals using a random effects model. Heterogeneity will be examined using the I2 statistic.

ELIGIBILITY:
Inclusion Criteria:

1. An aetiological healthy population study, the Whitehall II Study, comprising non-industrial civil servants aged 35-55 years who worked in the London offices of 20 civil service departments at baseline (1985-1988), will be used
2. A chest pain clinic cohort of consecutive ambulatory patients with no prior investigations for coronary disease and no prior history of acute coronary syndrome recruited in six rapid access chest pain clinics from 1996-2002
3. A coronary angiography cohort of consecutive patients undergoing elective angiography at three centres in London between 1996-1997
4. Patients with a record in MINAP between 1 Jan 2003 - latest date available in 2009. Only index MINAP events will be included in the analysis.

To obtain old data for meta-analysis, we will undertake a systematic review. We will search MEDLINE 1966-2008, without any language restriction, using relevant text words and search terms to find papers using the following inclusion criteria: coronary artery disease, South Asian ethnicity with White Caucasian comparison group, prospective study. We will use the MESH terms (India or Pakistan or Bangladesh or Sri Lanka or Ethnic Groups or ethnology or Asian Continental Ancestry Group or Asia) and (coronary or myocardial infarction or myocardial ischemia or cardiovascular disease). To focus further on longitudinal studies, the search will be expanded using a combination of all the Medline Clinical Queries filters for incidence and prognosis and including 'follow-up studies' and 'treatment/disease-outcome' as terms as well. The search will be repeated in Embase. Hand-searching of the reference list of eligible studies will be conducted to identify further relevant work (backward citation tracking). Science Citation Index will be used to identify all the subsequent papers that cited any of the eligible studies (forward citation tracking) using ISI Web of Science.

We will exclude any study that covers an ethnic group other than South Asian, studies not on coronary disease and studies that examined cross-sectional mortality or cross-sectional associations of cardiovascular risk factors with populations.

Exclusion Criteria:

admitted to hospital with fewer than 25 admissions in given year

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ACS registry data (MINAP) - with hospital admission databases (Hospital Episode Statistics (HES)
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 365 days
  365 days Mortality from all causes from the date of admission

SECONDARY OUTCOMES:
all causes in-hospital mortality | length of hospital stay
  death during duration of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Epidemiology Group, Department of Epidemiology & Public Health, UCL, London, United Kingdom

REFERENCES:
- [Derived] Zaman MJ, Philipson P, Chen R, Farag A, Shipley M, Marmot MG, Timmis AD, Hemingway H. South Asians and coronary disease: is there discordance between effects on incidence and prognosis? Heart. 2013 May;99(10):729-36. doi: 10.1136/heartjnl-2012-302925. Epub 2013 Feb 13. PMID 23406688